CLINICAL TRIAL: NCT00026793
Title: Protocol to Assess Vascularity in Kaposi's Sarcoma Lesions Utilizing Non-Invasive Imaging Techniques
Brief Title: Assessment of Blood Vessel Density in Kaposi's Sarcoma Lesions
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Yarchoan, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010158; 01-C-0158
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Kaposi's Sarcoma
Keywords: Kaposi Sarcoma; Doppler; Infrared; HIV; Imaging; Kaposi's Sarcoma; Laser Imaging; Infrared Imaging
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kaposi's Sarcoma: Adult patients with biopsy-proven cutaneous Kaposi's sarcoma. Some participants received interleukin-12 and liposomal doxorubicin. However, the therapy was administered on a different protocol and was not part of this study.

SUMMARY:
The purpose of this study is to develop imaging techniques to determine the density of blood vessels and the amount of blood flow in Kaposi s sarcoma (KS) tumors. KS tumors depend on the formation of new blood vessels for their growth. Some experimental therapies for KS are directed at reducing the amount of blood vessels and blood flow in these lesions. Measurement of blood vessel density and blood flow in these lesions could be useful in evaluating the effectiveness of both standard and experimental treatments for this disease.

Patients 18 years of age or older with Kaposi's sarcoma involving the skin may be eligible for this study. Participants will have photographs taken of their lesions and will undergo three imaging procedures (described below) at the beginning of the study (baseline) and then about once every 3 months or so while on the study (up to 2 years) to compare the test results over time. (Imaging may be done at more or less frequent intervals depending on the findings.) A small amount of blood (less than a tablespoon) will be drawn the day of each imaging procedure.

Laser Doppler imaging This technique measures the amount of blood flow in KS lesions by scanning the lesions with a low-power laser beam. Each lesion takes about 3 minutes to scan. The imaging may be done before and after a blood pressure cuff around the arm is inflated for a short time (usually less than 30 seconds).

Multi-spectral imaging This technique uses light to measure the total blood volume in each lesion and how much oxygen is in the blood. Oxygen is carried to the body s cells by a protein in red blood cells called hemoglobin. The light on the multi-spectral imaging instrument is absorbed differently depending on whether the hemoglobin has oxygen attached to it or not. It takes about 2 minutes to scan each lesion.

Infrared thermal imaging This test uses a special camera to take digital infrared pictures of the skin. Images formed of the temperature of the KS lesions are used to assess blood flow in the lesions. This imaging takes about 1 minute per lesion.

...

DETAILED DESCRIPTION:
Background:

Kaposi's sarcoma is a highly vascular tumor. As such, it may provide a good model for the study of angiogenesis-based therapy in cancer. However, there are no standardized techniques now available to assess the effects of anti-angiogenesis therapy on blood flow in KS tissues. The present protocol was written to allow us to explore and gain experience with four promising techniques to examine tumor vasculature in cutaneous KS lesions: a) laser Doppler imaging; b) multi-spectral imaging; c) infrared thermal imaging; and d) optical coherence tomography.

Objectives:

The main objective is to assess, in preliminary fashion, non-invasive methods for studying tumor vascularity and vascular changes in patients with Kaposi's sarcoma using four different imaging techniques. Other objectives are to correlate these techniques to each other and to conventional KS tumor assessment, and to assess the response of these techniques in patients receiving therapy for Kaposi s sarcoma.

Eligibility:

Patients 18 of more years of age with biopsy-proven cutaneous Kaposi's sarcoma involving the skin or mucosa are eligible. They must be willing and able to give informed consent.

Design:

This will be a preliminary study to explore these techniques in Kaposi's sarcoma. Selected Kaposi's sarcoma lesions of patients will be assessed using laser Doppler imaging, multi-spectral imaging, infrared thermal imaging, and optical coherence tomography at entry and then additional time points for up to 4 years. Lesions will also be assessed by conventional measurement and photographs with conventional cameras. In selected patients in which there are Kaposi's sarcoma lesions on the arm, the effects of stopping venous flow for up to 10 seconds will be assessed on the measurements. A complete blood count will be done the day of the measurements. The results of the imaging techniques will be compared with each other, and with conventional tumor assessments. Changes over time will be assessed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Biopsy proven Kaposi's sarcoma involving the skin or mucosa.

Age greater than or equal to 18 years.

EXCLUSION CRITERIA:

Unable or unwilling to give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject selection will primarily be from patients with Kaposi's Sarcoma enrolled on other protocols in the human immunodeficiency virus (HIV) and Acquired immunodeficiency syndrome (AIDS) Malignancy Branch. Other sources will be referrals from other institutes and physicians.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2001-04-23 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ensoli B, Nakamura S, Salahuddin SZ, Biberfeld P, Larsson L, Beaver B, Wong-Staal F, Gallo RC. AIDS-Kaposi's sarcoma-derived cells express cytokines with autocrine and paracrine growth effects. Science. 1989 Jan 13;243(4888):223-6. doi: 10.1126/science.2643161.
- [Background] Miles SA, Rezai AR, Salazar-Gonzalez JF, Vander Meyden M, Stevens RH, Logan DM, Mitsuyasu RT, Taga T, Hirano T, Kishimoto T, et al. AIDS Kaposi sarcoma-derived cells produce and respond to interleukin 6. Proc Natl Acad Sci U S A. 1990 Jun;87(11):4068-72. doi: 10.1073/pnas.87.11.4068. PMID 1693429
- [Background] Friedlander M, Brooks PC, Shaffer RW, Kincaid CM, Varner JA, Cheresh DA. Definition of two angiogenic pathways by distinct alpha v integrins. Science. 1995 Dec 1;270(5241):1500-2. doi: 10.1126/science.270.5241.1500. PMID 7491498
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2001-C-0158.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kaposi's Sarcoma
Started | 29
Completed | 21
Not Completed | 8
Not completed — Death on study due to underlying disease | 4
Not completed — Physician Decision | 2
Not completed — Off study | 2

BASELINE CHARACTERISTICS:
Groups:
- Kaposi's Sarcoma: Adult patients with biopsy-proven cutaneous Kaposi's sarcoma
Arm/Group | Kaposi's Sarcoma
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.69 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 15
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Preliminary Assessment of the Temperature of Kaposi's Sarcoma Lesions Compared to the Temperature in the Normal Skin Measured With Thermography
Description: Temperature in KS lesions compared to normal skin either adjacent to the lesion or on the contralateral side was measured with thermography (thermal energy). A higher temperature is proportional to the severity of the lesion (worst outcome). A reduction in temperature is consistent with a decrease in severity of the lesions (better outcome).
Time Frame: Baseline (prior to therapy)
Population: Only 16/29 participants were analyzed for this outcome measure. Due to the assay being developed, results data were not collected in a consistent manner for the remaining 13 participants.
Measure: Median (Full Range); unit: Celsius
Arm/Group | Kaposi's Sarcoma
Number analyzed (Participants) | 16
Celsius | 1.1 [-0.68 to 3.43]

2. Secondary Outcome: Preliminary Assessment of the Blood Velocity in Kaposi's Sarcoma (KS) Lesions Compared to That in the Surrounding Area
Description: Blood velocity in Kaposi's Sarcoma lesions as compared to the surrounding area was measured with laser doppler imaging with a low power laser beam. Higher velocity is an indication of more severe lesions.
Time Frame: Baseline (prior to therapy)
Population: as for outcome 1
Measure: Median (Full Range); unit: Arbritary units (AU)
Arm/Group | Kaposi's Sarcoma
Number analyzed (Participants) | 16
Arbritary units (AU) | 66 [-44 to 451]

3. Secondary Outcome: Preliminary Assessment of the Temperature Change in Kaposi Sarcoma Lesions at Week 18 of Therapy Compared to Baseline as Measured With Thermography
Description: Temperature in KS lesions compared to normal skin either adjacent to the lesion or on the contralateral side was measured with thermography (thermal energy). A higher temperature is proportional to the severity of the lesion (worst outcome). A reduction in temperature is consistent with a decrease in severity of the lesions (better outcome). The value at week 18 is compared to the baseline value for each subject, and the difference reported.
Time Frame: Baseline and 18 weeks after therapy
Population: Only 10/29 participants were analyzed for this outcome measure.
Measure: Median (Full Range); unit: Celsius
Arm/Group | Kaposi's Sarcoma
Number analyzed (Participants) | 10
Celsius | -0.985 [-2.99 to 0.4]

4. Secondary Outcome: Preliminary Assessment of the Change in Blood Velocity in Kaposi's Sarcoma Lesions Measured With Laser Doppler Imaging Before and After Therapy
Description: Blood velocity in Kaposi's Sarcoma lesions as compared to the surrounding area was measured with laser doppler imaging with a low power laser beam. Higher velocity is an indication of more severe lesions. The value at week 18 is compared to the baseline value for each subject, and the difference reported.
Time Frame: Baseline and 18 weeks after therapy
Population: Only 10/29 participants were analyzed for this outcome measure.
Measure: Median (Full Range); unit: Change in arbritary units (AU)
Arm/Group | Kaposi's Sarcoma
Number analyzed (Participants) | 10
Change in arbritary units (AU) | -115 [-305 to -17]

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 196 months and 19 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Kaposi's Sarcoma
Number analyzed (Participants) | 29
Participants | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 196 months and 19 days.
Arm/Group | Kaposi's Sarcoma
All-Cause Mortality (participants affected / at risk) | 4/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-21): https://cdn.clinicaltrials.gov/large-docs/93/NCT00026793/Prot_SAP_000.pdf
  • Informed Consent Form (2013-11-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT00026793/ICF_001.pdf